CLINICAL TRIAL: NCT05781789
Title: Redesigning Pre-surgery Patient Journeys With Telehealth
Status: Active, not recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Nanyang Technological University (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: AM/HRT/008/2021
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Surgery
Keywords: Preoperative evaluation; Telehealth
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient participants: Patient booked for elective surgery and:
  Age 21 to 70 years English literacy Willing to provide signed consent Of any nationality Able to give own legal consent
  Interventions: Other: Telehealth for preoperative evaluation
- Healthcare provider participants: Criteria:
  * Age 21 to 70 years
  * Healthcare professionals comprising clinic staff (surgical outpatient clinics, PAS), clinicians (anaesthetists, surgeons), and health service managers)
  * working in the perioperative clinical areas
  Interventions: Other: Telehealth for preoperative evaluation

INTERVENTIONS:
Other: Telehealth for preoperative evaluation — Conduct of preoperative evaluation remotely using Zoom application
  Other Names: Video consultation

SUMMARY:
Prior to surgery, patients undergo preanaesthesia assessment to ensure timely optimisation of medical conditions that could adversely impact perioperative outcomes. At the Preadmission Service (PAS) clinic of KK hospital, nurses perform the first triage to identify patients who require outpatient anaesthetic review in advance of surgery. While all elective patients attend the PAS clinic, only 8% are require outpatient anaesthetic review. The majority 92%, can be safely triaged to receive preanaesthesia assessment on the day of surgery. In this project, the investigators propose to investigate the efficacy of a new pre-surgery workflow for elective surgical patients incorporating telehealth. The investigators hypothesize that the redesigned pre-surgery journey incorporating telehealth reduces in-person consultation at the pre-admission clinic by up to 90%. Primary outcome is the proportion of eligible same-day-admission patients assessed via telehealth. Secondary outcomes are:

1. Patient cost and time savings
2. Patient experience of the new model of care
3. Staff experience of the new workflow
4. Incidence of day-of-surgery cancellations

DETAILED DESCRIPTION:
Prior to elective surgery, patients undergo preanaesthesia assessment to ensure timely optimisation of medical conditions that could adversely impact perioperative outcomes. Preadmission Service (PAS) clinic nurses at KK Hospital perform pre-surgery triage to identify patients requiring outpatient anaesthetic review. PAS data shows that only 8% of same-day-admission (SDA) patients needed an anaesthetist's review; the majority (92%) can be safely triaged to receive preanaesthesia assessment on the day of surgery. The aim of this study is to investigate the service re-design, efficacy and effectiveness of a new telehealth pre-surgery model of care for elective SDA patients. The investigators hypothesize that the telehealth pre-surgery new model of care will achieve an expected 50% uptake for SDA patients as the primary outcome during implementation. Secondary outcomes are patient cost savings, patient experience of the new model of care, and staff experience of the new workflow. The investigators will use a sequential exploratory mixed methods study design, consistent with the 5-stage model for telehealth research. An implementation science framework - the Normalisation Process Theory, underpins our 3-phase study. Phase 1 (service redesign) explores the feasibility of presrugery telehealth via semi-structured interviews of patients and healthcare staff. Phase 2 (preimplementation) investigates efficacy of the telehealth model of care by addressing service fidelity, and patient and staff experience using administrative data. Phase 3 is a pragmatic trial to ascertain effectiveness of the telehealthmodel of care, addressing the primary and secondary outcomes stated. This novel study using implementation science to redesign and implement presurgery telehealth will inform scale-up, spread, and sustainability of a new model of care within SingHealth and other health clusters in Singapore.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants:

Age 21 to 70 years Listed for elective surgery English literacy Willing to provide signed consent Of any nationality Able to give own legal consent

Exclusion Criteria:

* Healthcare participants:

Age 21 to 70 years Healthcare professionals comprising clinic staff (surgical outpatient clinics, PAS), clinicians (anaesthetists, surgeons), and health service managers)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patient participants are female as they are recruited from a women's hospital
Study Population: Patient participants are female patients booked for elective surgery at a tertiary women's hospital.
  Healthcare participants are nurses, administrators, surgeons and anaesthetists working in the preoperative and surgeons' clinics at a tertiary women's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible elective surgery patients assessed successfully via telehealth for preoperative evaluation | One year from the initiation of the implementation phase (Phase 3)
  Of the total number of patients booked for elective surgery, the proportion of patients evaluated preoperatively by telehealth is measured.

SECONDARY OUTCOMES:
Patient's perception and attitude towards a Telehealth model of care for preoperative evaluation | 5 months from July to November 2021
  Quantitative study via one-on-one semi-structured interviews of elective surgery patients to evaluate their attitudes and perception of the new proposed telehealth workflow conducted in (Service Redesign) Phase 1
Healthcare providers' perception and attitude towards a Telehealth model of care for preoperative evaluation | 5 months from July to November 2021
  Quantitative study via one-on-one semi-structured interviews of healthcare providers working in the peroperative and surgery clinics to evaluate their attitudes and perception of the new proposed telehealth workflow conducted in (Service Redesign) Phase 1

CONTACTS AND LOCATIONS:
Overall Officials: Chai-Rick Soh, FANZCA, Study Chair — Singapore General Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wong DT, Kamming D, Salenieks ME, Go K, Kohm C, Chung F. Preadmission anesthesia consultation using telemedicine technology: a pilot study. Anesthesiology. 2004 Jun;100(6):1605-7. doi: 10.1097/00000542-200406000-00038. No abstract available. PMID 15166585
- [Result] Applegate RL 2nd, Gildea B, Patchin R, Rook JL, Wolford B, Nyirady J, Dawes TA, Faltys J, Ramsingh DS, Stier G. Telemedicine pre-anesthesia evaluation: a randomized pilot trial. Telemed J E Health. 2013 Mar;19(3):211-6. doi: 10.1089/tmj.2012.0132. Epub 2013 Feb 5. PMID 23384334
- [Result] Mullen-Fortino M, Rising KL, Duckworth J, Gwynn V, Sites FD, Hollander JE. Presurgical Assessment Using Telemedicine Technology: Impact on Efficiency, Effectiveness, and Patient Experience of Care. Telemed J E Health. 2019 Feb;25(2):137-142. doi: 10.1089/tmj.2017.0133. Epub 2018 Jul 26. PMID 30048210
- [Result] Murray E, Treweek S, Pope C, MacFarlane A, Ballini L, Dowrick C, Finch T, Kennedy A, Mair F, O'Donnell C, Ong BN, Rapley T, Rogers A, May C. Normalisation process theory: a framework for developing, evaluating and implementing complex interventions. BMC Med. 2010 Oct 20;8:63. doi: 10.1186/1741-7015-8-63. PMID 20961442
- [Result] Donelan K, Barreto EA, Sossong S, Michael C, Estrada JJ, Cohen AB, Wozniak J, Schwamm LH. Patient and clinician experiences with telehealth for patient follow-up care. Am J Manag Care. 2019 Jan;25(1):40-44. PMID 30667610
- [Derived] Lew E, Tan SFJ, Teo A, Sng BL, Lum EPM. Perceptions and Attitudes of Patients and Health Care Stakeholders on Implementing a Telehealth Service for Preoperative Evaluation: A Qualitative Analysis. Telemed Rep. 2023 Jun 26;4(1):156-165. doi: 10.1089/tmr.2023.0023. eCollection 2023. PMID 37771697